CLINICAL TRIAL: NCT01920724
Title: Body Composition and Dietary Intake in Preschool Children Aged 3-5 Years in Daycare Centers
Brief Title: Body Composition in Preschool Children
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: MU-IRB 2010/211.0807; A09/2554 (Other Grant/Funding Number: Mahidol University)
Record Dates: First submitted 2013-07-13; First posted 2013-08-12 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Wasting
Keywords: Preschool children; Body composition
MeSH Terms: conditions — Obesity; Cachexia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- wasting, obesity, stunting, normal: wasting (BMI for age Z-scores < -2 SD), normal (-1 SD ≤ BMI for age Z-scores ≤ +1 SD), obesity (BMI for age Z-scores > +2 SD), and stunting (HAZ < -2 SD).

SUMMARY:
Thailand has been facing with the double burden of malnutrition. Many studies in Thailand, which aim to explore the situation, causes, and strategies to prevent obesity, have focused on adults, adolescents, or school-aged children. Few studies have been conducted in preschool children. Obesity or stunting during childhood increases the risk of being obesity in adulthood and leads to chronic diseases. If obesity is established in adulthood, it is difficult to reduce the excess weight. Thus, the prevention of obesity or stunting in young children should be highly considered. Study of dietary pattern and reliable field methods to measure fat mass (FM) in children may partly contribute to primary prevention of childhood obesity. The deuterium dilution technique is an accurate and suitable method for children and population-based studies. However, it has not been widely used in children in Thailand. Hence, this study aimed to utilize the deuterium dilution technique for assessing body composition and to determine the quality and quantity of dietary intake among children 3-5 years of age with different nutritional status. We conducted a cross-sectional study in 15 daycare centers in Nakhon Pathom and Samut Prakarn provinces. 120 preschoolers were purposively selected according to their nutritional status: stunted, thin, normal, and overweight/obese. Anthropometric measurements were conducted. Body composition was determined based on total body water using deuterium dilution technique. Dietary intake data were obtained using 2-day 24 hr recall.We hypothesized that stunted and obese children will have more fat mass compared to the normal children.

DETAILED DESCRIPTION:
Body composition of the children was assessed using the deuterium technique. Total body water (TBW) content was calculated. Then, fat free mass (FFM) and fat mass (FM) was calculated.

Weight and height of all children were using a standard technique. Body mass index and nutritional status was calculated using World Health Organization (WHO) growth standard for children 0-5 years.

Dietary intake of children was assessed using 2 non-consecutive 24 hour dietary recalls. The 1st and 2nd recall was about 2 weeks apart. Nutrient intake was calculated using the INMUCAL-Nutrients WD. 4.0 (Institute of Nutrition, 2010).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Aged 3-5 years
* BMI or HAZ fall in the study protocol

Exclusion Criteria:

* Chronic diseases
* Ongoing medical treatments likely to affect body composition
* Malformation or muscle diseases

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in the daycare centers in Nakhon Pathom and Samut Prakarn porvinces will be screened and categorized into 4 groups, including wasting (BMI for age Z-scores < -2 SD), normal (-1 SD ≤ BMI for age Z-scores ≤ +1 SD), obesity (BMI for age Z-scores > +2 SD), and stunting (HAZ < -2 SD). Then, they will be randomly selected to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Body composition | 4 months
  Body fatness

SECONDARY OUTCOMES:
Nutrient intake | 4 months
  24 hr recall was perform on a weekend day and a weekday day and nutrient intake was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Institute of Nutrition, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Introduction to body composition assessment — http://www-pub.iaea.org/MTCD/publications/PDF/Pub1451_web.pdf